CLINICAL TRIAL: NCT02662530
Title: Comparison of Clinical and Kinematic Assessment in the Determination of Botox® Injection Parameters in Cervical Dystonia Patients
Brief Title: Clinical and Kinematic Assessment for Determination of Botox® Injection Parameters in Cervical Dystonia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Mandar Jog, Principal Investigator, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 105515
Record Dates: First submitted 2016-01-07; First posted 2016-01-25 (Estimated); Last update posted 2020-06-22 (Actual); Status verified 2020-06

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum toxin type A clinical (Active Comparator): Initial and optimization of BoNT-A injection parameters will be conducted by clinical visual assessment
  Interventions: Drug: Botulinum Toxin Type A
- Botulinum toxin type A kinematic (Active Comparator): Initial and optimization of BoNT-A injection parameters will be conducted by kinematic assessment
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Drug: Botulinum Toxin Type A — A serotype of botulinum toxin type A (BoNT-A) that has specificity for cleavage of SYNAPTOSOMAL-ASSOCIATED PROTEIN 25 (SNAP-25). BoNT-A's pharmacological action is to inhibit the release of acetylcholine from the neuromuscular junction. BoNT-A peripherally applied using optimal parameters by intramuscular injections solely determined either by visual/clinical or by biomechanical analysis of dystonic movements for cervical dystonia therapy in neck and shoulder muscles every 12 weeks over 30 weeks. BoNT-A dose will range from 50-300 U.
  Other Names: Botox; onabotulinumtoxinA

SUMMARY:
This study investigates the use of a kinematic measurement device to quantify the abnormal head movements and postures in patients with cervical dystonia (CD) in order to individualize and optimize botulinum toxin type A (BoNT-A) injection therapy. A single sensor captures five degrees of freedom of the neck and head that distinguish which muscle(s) contribute to CD and the amount of BoNT-A to inject into these muscle(s). The efficacy, relief and improvements in social, occupation and function by injections will be investigated. The efficacy of BoNT-A therapy using either BoNT-A injection parameters from clinical-based assessments and kinematically-based assessments will be investigated in CD patients. Individuals clinically diagnosed with CD will be randomized for two treatment conditions: A) injection parameters from a kinematic assessment only, or B) injection parameters from a clinical assessment only.

ELIGIBILITY:
Inclusion Criteria:

* Consenting male and female individuals between the ages of 18 and 80
* Diagnosed with idiopathic spasmodic torticollis (also called cervical dystonia) by neurologist
* Botulinum neurotoxin type A injection(BoNT A; Botox®) naïve individuals will be randomized into either clinical-assessment arm or kinematic-assessment arm and the participants will be blinded to which arm they are a part of
* CD individuals who are receiving suboptimal BoNT-A effects will be recruited to receive kinematic-based injections. These participants will have to wait a minimum of 4 months before participating in this study
* Able to attend all study sessions
* Able to provide written consent

Exclusion Criteria:

* Pregnant individuals
* Women who are nursing
* Individuals with a known Botox® allergy
* Individuals with a known or suspected traumatic cause for the torticollis, a prior thalamotomy, or peripheral (nerve or muscle) operation
* Individuals with cervical contractures that limit passive range of motion
* Motor/nerve diseases such as myasthenia gravis, other diseases of the neuromuscular junction and/or Amyotrophic Lateral Sclerosis
* Myotomy or denervation surgery involving the neck or shoulder region

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with significant relief of severity and pain by TWSTRS part A and C, respectively, over treatment course | 30 weeks
  Physiological changes as a result of BoNT-A injection treatment will be assessed by validated CD assessment scale, TWSTRS part A for severity and C for pain, will be administered at each time-point to determine efficacy of using BoNT-A parameters based on clinical versus kinematics.
Number of participants with significant relief of severity by objective kinematic reductions in angular deviation and amplitude measures over treatment course | 30 weeks
  Number of participants with significant relief of severity by objective kinematic reductions in angular deviation and amplitude measures over treatment course. Physiological changes in static/natural neck and head posturing, dynamic/tremor/dystonic movements superimposed on natural head position, range of motion will be assessed kinematically at each time-point. Angular deviations are calculated by degree of freedom angular bias from calibrated neutral position. Amplitude measures will be reported as root mean square values.

SECONDARY OUTCOMES:
Number of participants with significant improvement in functional disability scores assessed by TWSTRS part B and patient-reported scores pre- and post-BoNT-A parameters determined visually or kinematically. | 30 weeks
  Change in functional disability, quality of life and relief of pain as a result of BoNT-A injection treatment will be measured will be measured by comparing pre- and post-injection TWSTRS.
Number of participants with significant relief of severity by global impression of change scores over treatment course | 30 weeks
  Number of participants with significant relief of severity and pain by global impression of change scores over treatment course. This scale is a self-reported by participant on a VAS/Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Mandar Jog, MD, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Brans JW, Lindeboom R, Snoek JW, Zwarts MJ, van Weerden TW, Brunt ER, van Hilten JJ, van der Kamp W, Prins MH, Speelman JD. Botulinum toxin versus trihexyphenidyl in cervical dystonia: a prospective, randomized, double-blind controlled trial. Neurology. 1996 Apr;46(4):1066-72. doi: 10.1212/wnl.46.4.1066. PMID 8780093
- [Background] Caleo M, Antonucci F, Restani L, Mazzocchio R. A reappraisal of the central effects of botulinum neurotoxin type A: by what mechanism? J Neurochem. 2009 Apr;109(1):15-24. doi: 10.1111/j.1471-4159.2009.05887.x. Epub 2009 Feb 11. PMID 19154335
- [Background] Dressler D. Botulinum toxin for treatment of dystonia. Eur J Neurol. 2010 Jul;17 Suppl 1:88-96. doi: 10.1111/j.1468-1331.2010.03058.x. PMID 20590814
- [Background] Evidente VG, Truong D, Jankovic J, Comella CL, Grafe S, Hanschmann A. IncobotulinumtoxinA (Xeomin(R)) injected for blepharospasm or cervical dystonia according to patient needs is well tolerated. J Neurol Sci. 2014 Nov 15;346(1-2):116-20. doi: 10.1016/j.jns.2014.08.004. Epub 2014 Aug 10. PMID 25186131
- [Background] Evidente VG, Pappert EJ. Botulinum toxin therapy for cervical dystonia: the science of dosing. Tremor Other Hyperkinet Mov (N Y). 2014 Nov 12;4:273. doi: 10.7916/D84X56BF. eCollection 2014. PMID 25414799
- [Background] Werdelin L, Dalager T, Fuglsang-Frederiksen A, Regeur L, Karlsborg M, Korbo L, Munck O, Winge K. The utility of EMG interference pattern analysis in botulinum toxin treatment of torticollis: a randomised, controlled and blinded study. Clin Neurophysiol. 2011 Nov;122(11):2305-9. doi: 10.1016/j.clinph.2011.04.012. Epub 2011 Jun 1. PMID 21636319
- [Background] Raez MB, Hussain MS, Mohd-Yasin F. Techniques of EMG signal analysis: detection, processing, classification and applications. Biol Proced Online. 2006;8:11-35. doi: 10.1251/bpo115. Epub 2006 Mar 23. PMID 16799694